CLINICAL TRIAL: NCT03733210
Title: Pilot Study Evaluating Panitumumab-IRDye800 and 89Zr-Panitumumab for Dual-Modality Imaging for Nodal Staging in Head and Neck Cancer
Brief Title: Panitumumab-IRDye800 and 89Zr-Panitumumab in Identifying Metastatic Lymph Nodes in Patients With Squamous Cell Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-41878; NCI-2018-02270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ENT0066 (Other: OnCore Number); P30CA124435 (NIH); R01CA190306 (NIH)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Carcinoma of the Head and Neck
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tumor-negative Lymph Nodes (by 18F-FDG scan) (Experimental): Participants whose lymph nodes are negative for cancer
  Interventions: Drug: Panitumumab-IRDye800; Drug: 89-Zirconium (Zr-89) Panitumumab; Device: Pinpoint IR IR9000 fluorescence imaging system (FIS); Device: SPY-PHI IR9000 fluorescence imaging system (FIS); Device: Explorer Air camera; Device: PDE-NEO II camera; Device: FIS-00 fluorescence imaging system (FIS); Device: Da Vinci Firefly Imaging System; Device: IGP-ELVIS-v4 Macroscopic Specimen Imager; Device: Vevo 3100 LAZR-X; Device: Pearl Triology Imaging System; Device: Odyssey CLx Imaging System; Device: Leica fluorescence microscope
- Tumor-positive Lymph Nodes (by 18F-FDG scan) (Experimental): Participants whose lymph nodes are positive for cancer.
  Interventions: Drug: Panitumumab-IRDye800; Drug: 89-Zirconium (Zr-89) Panitumumab; Device: Pinpoint IR IR9000 fluorescence imaging system (FIS); Device: SPY-PHI IR9000 fluorescence imaging system (FIS); Device: Explorer Air camera; Device: PDE-NEO II camera; Device: FIS-00 fluorescence imaging system (FIS); Device: Da Vinci Firefly Imaging System; Device: IGP-ELVIS-v4 Macroscopic Specimen Imager; Device: Vevo 3100 LAZR-X; Device: Pearl Triology Imaging System; Device: Odyssey CLx Imaging System; Device: Leica fluorescence microscope

INTERVENTIONS:
Drug: Panitumumab-IRDye800 — 30 mg administered intravenously (IV)
  Other Names: Panitumumab IRDye 800; IRDye800-Panitumumab Conjugate
Drug: 89-Zirconium (Zr-89) Panitumumab — 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Other Names: 89Zr-panitumumab (SY); 89Zr-labeled Panitumumab (SY); Zr 89-Panitumumab (SY)
Device: Pinpoint IR IR9000 fluorescence imaging system (FIS) — Handheld fluorescence-imaging endoscope manufactured by Novadaq
Device: SPY-PHI IR9000 fluorescence imaging system (FIS) — Handheld fluorescence-imaging endoscope manufactured by Novadaq
Device: Explorer Air camera — Fluorescence camera manufactured by SurgVision
Device: PDE-NEO II camera — Medical infrared camera manufactured by Hamamatsu Photonics KK
Device: FIS-00 fluorescence imaging system (FIS) — Fluorescence-imaging system (FIS) manufactured by Hamamatsu Photonics KK
Device: Da Vinci Firefly Imaging System — Fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
Device: IGP-ELVIS-v4 Macroscopic Specimen Imager — Macroscopic specimen imager manufactured by LI-COR Biosciences
Device: Vevo 3100 LAZR-X — Photoacoustic ultrasound imaging system manufactured by VisualSonics
Device: Pearl Triology Imaging System — Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
Device: Odyssey CLx Imaging System — Infrared fluorescent-imaging system manufactured by LI-COR Biosciences
Device: Leica fluorescence microscope — Fluorescence microscope manufactured by Leica

SUMMARY:
This study evaluates how well panitumumab-IRDye800 and 89Zr-panitumumab work in identifying cancer that has spread to the lymph nodes in patients with squamous cell head and neck cancer. Panitumumab-IRDye800 is a drug that contains a dye molecule that fluoresces during surgery to indicate cancerous tissue. 89Zr-panitumumab is a drug that contains a small amount of radiation, which makes it visible in positron emission tomography (PET) scans. PET scans make detailed, computerized pictures of areas inside the body where the drug is used. Giving panitumumab-IRDye800 and 89Zr-panitumumab to patients with head and neck cancer may help doctors find metastatic lymph nodes better than current methods [positron emission tomography (PET); computed tomography (CT); magnetic imaging resonance (MRI), or combinations].

DETAILED DESCRIPTION:
For patients with head and neck cancer, detection of malignant cells within nearby lymph nodes (LNs) is an important measure of the extent and severity of the cancer. LNs are a key immunologic organ involved in overall immune surveillance. Historically, LN or LNs were harvested before the surgery of curative intent, evaluated pathologically, and then tumor status of the harvested LNs were utilized to inform the individual surgical plan. These LNs became known as "sentinel lymph nodes." In recent years, techniques have been developed to utilize peritumoral injection (around the tumor) of tumor labels that could identify tumor in the LNs without biopsy, ie, only LNs that were tumor-positive would be removed. However, in some patients, this technique could be limited by the location of the primary cancer. Effective and sensitive systemically-administered labels would be a significant advancement. The systemically-administered label 18F-fluorodeoxyglucose (18F-FDG), detected by positron emission tomography / computed tomography (PET/CT) and/or PET / magnetic imaging resonance (PET/MRI) radiologic scans and representing current regular medical care, has provided improvement in detection of cancer-positive LNs. However, further enhancements may be possible.

Participants with squamous cell carcinoma of the head and neck (SCCHN) and scheduled to undergo regular medical care surgery with curative intent, were assigned to 2 study groups on the basis of whether regular medical care scans using 18F-FDG PET/CT or PET/MRI had indicated that cancer was suspected in the lymph nodes (LN+ or cN+), or without suspected cancer in the lymph nodes (LN- or cN0). Following the 18F-FDG, and prior to surgery, 89Zr-panitumumab was systemically administered by intravenous infusion, and a PET-CT imaging scan was conducted. Research imaging will be performed intraoperatively using optical imaging devices and a high-energy gamma probe. Subsequently, the excised tissue will evaluated ex vivo (back table) using radioactive (89Zr-panitumumab) and fluorescence (panitumumab-IRDye800) imaging techniques. Regular medical care surgical excision of the tumor and adjacent LN was conducted on Day 2 to 5. After surgery, patients are followed up at 15 and 30 days.

PRIMARY OBJECTIVES:

I. Determine the sensitivity and specificity of zirconium(89Zr)-panitumumab (89Zr-panitumumab) for the detection of tumor-involved regional lymph nodes.

SECONDARY OBJECTIVES:

I. Determine the number (proportion) of lymph nodes determined to be tumor positive by histological and/or pathological evaluation that were NOT predicted tumor-positive by 89Zr-panitumumab labeling.

EXPLORATORY OBJECTIVES:

I. Determine the sensitivity and specificity of panitumumab-IRDye800 for the detection of tumor-involved regional lymph nodes.

II. Determine the number (proportion) of lymph nodes determined to be tumor positive by histological and/or pathological evaluation that were NOT predicted tumor-positive by panitumumab-IRDye800 labeling.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck.
* Subjects diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Subjects with recurrent disease or a new primary will be allowed.
* Planned standard of care surgery with curative intent for squamous cell carcinoma.
* Hemoglobin ≥ 9 gm/dL.
* White blood cell count > 3000/mm³.
* Platelet count ≥ 100,000/mm³.
* Serum creatinine ≤ 1.5 times upper reference range.

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
* Previous bilateral neck dissection.
* History of infusion reactions to monoclonal antibody therapies.
* Pregnant or breastfeeding.
* Magnesium or potassium lower than the normal institutional values.
* Subjects receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
* Severe renal disease or anuria.
* Known hypersensitivity to deferoxamine or any of its components.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford Medicine at Stanford University
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tumor-negative Lymph Nodes (by 18F-FDG Scan): Participants whose lymph nodes are negative for cancer
  Panitumumab-IRDye800: 30 mg administered intravenously (IV)
  Zirconium Zr-89 Panitumumab: 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Pinpoint IR IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  SPY-PHI IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  Explorer Air camera: Fluorescence camera manufactured by SurgVision
  PDE-NEO II camera: Medical infrared camera manufactured by Hamamatsu Photonics KK
  FIS-00 fluorescence imaging system (FIS): Fluorescence imaging system (FIS) manufactured by Hamamatsu Photonics KK
  Da Vinci Firefly Imaging System: Fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
  IGP-ELVIS-v4 Macroscopic Specimen Imager: Macroscopic specimen imager manufactured by LI-COR Biosciences
  Vevo 3100 LAZR-X: Photoacoustic ultrasound imaging system manufactured by VisualSonics
  Pearl Triology Imaging System: Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
  Odyssey CLx Imaging System: Infrared fluorescent imaging system manufactured by LI-COR Biosciences
  Leica fluorescence microscope: Fluorescence microscope manufactured by Leica
- Tumor-positive Lymph Nodes (by 18F-FDG Scan): Participants whose lymph nodes are positive for cancer.
  Panitumumab-IRDye800: 30 mg administered intravenously (IV)
  Zirconium Zr-89 Panitumumab: 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Pinpoint IR IR9000 fluorescence imaging system (FIS): Handheld fluorescence -imaging endoscope manufactured by Novadaq
  SPY-PHI IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  Explorer Air camera: Fluorescence camera manufactured by SurgVision
  PDE-NEO II camera: Medical infrared camera manufactured by Hamamatsu Photonics KK
  FIS-00 fluorescence imaging system (FIS): Fluorescence imaging system (FIS) manufactured by Hamamatsu Photonics KK
  Da Vinci Firefly Imaging System: fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
  IGP-ELVIS-v4 Macroscopic Specimen Imager: Macroscopic specimen imager manufactured by LI-COR Biosciences
  Vevo 3100 LAZR-X: Photoacoustic ultrasound imaging system manufactured by VisualSonics
  Pearl Triology Imaging System: Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
  Odyssey CLx Imaging System: Infrared fluorescent imaging system manufactured by LI-COR Biosciences
  Leica fluorescence microscope: Fluorescence microscope manufactured by Leica
Period: Overall Study
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
Started | 7 | 7
Completed | 3 | 5
Not Completed | 4 | 2
Not completed — Lymph nodes not collected or not evaluable | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Tumor-negative Lymph Nodes (by 18F-FDG Scan): Participants whose lymph nodes are negative for cancer
  Panitumumab-IRDye800: 30 mg administered intravenously (IV)
  Zirconium Zr-89 Panitumumab: 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Pinpoint IR IR9000 fluorescence-imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  SPY-PHI IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  Explorer Air camera: Fluorescence camera manufactured by SurgVision
  PDE-NEO II camera: Medical infrared camera manufactured by Hamamatsu Photonics KK
  FIS-00 fluorescence imaging system (FIS): Fluorescence-imaging system (FIS) manufactured by Hamamatsu Photonics KK
  Da Vinci Firefly Imaging System: Fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
  IGP-ELVIS-v4 Macroscopic Specimen Imager: Macroscopic specimen imager manufactured by LI-COR Biosciences
  Vevo 3100 LAZR-X: Photoacoustic ultrasound imaging system manufactured by VisualSonics
  Pearl Triology Imaging System: Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
  Odyssey CLx Imaging System: Infrared fluorescent imaging system manufactured by LI-COR Biosciences
  Leica fluorescence microscope: Fluorescence microscope manufactured by Leica
- Tumor-positive Lymph Nodes (by 18F-FDG Scan): Participants whose lymph nodes are positive for cancer.
  Panitumumab-IRDye800: 30 mg administered intravenously (IV)
  Zirconium Zr-89 Panitumumab: 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Pinpoint IR IR9000 fluorescence-imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  SPY-PHI IR9000 fluorescence-imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  Explorer Air camera: Fluorescence camera manufactured by SurgVision
  PDE-NEO II camera: Medical infrared camera manufactured by Hamamatsu Photonics KK
  FIS-00 fluorescence imaging system (FIS): Fluorescenc3-imaging system (FIS) manufactured by Hamamatsu Photonics KK
  Da Vinci Firefly Imaging System: Fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
  IGP-ELVIS-v4 Macroscopic Specimen Imager: Macroscopic specimen imager manufactured by LI-COR Biosciences
  Vevo 3100 LAZR-X: Photoacoustic ultrasound imaging system manufactured by VisualSonics
  Pearl Triology Imaging System: Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
  Odyssey CLx Imaging System: Infrared fluorescent imaging system manufactured by LI-COR Biosciences
  Leica fluorescence microscope: Fluorescence microscope manufactured by Leica
- Total: Total of all reporting groups
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 63.8 [56.2 to 79.8] | 69.8 [54.6 to 83.7] | 68.3 [54.6 to 83.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Detection of Tumor in Lymph Nodes by 18F-FDG and 89Zr-panitumumab Labeling
Description: The ability of 89Zr-panitumumab and 18F-fluorodeoxyglucose (18F-FDG) to detect tumor in lymph nodes were assessed on the basis of radiologic scans and histopathologic evaluation of excised lymph nodes (LNs). The histopathologic assessment was considered the definitive, regular medical care, assessment. The outcome is reported by study group as the number of LNs that were identified as tumor-positive by 18F-FDG- and 89Zr-panitumumab, stratified by the tumor-positivity as assessed by histopathology, and expressed as the number of LNs that were tumor-positive by both, negative for both, or positive for one and not the other. Results are also provided by study group for the number of LNs that tumor-positive by both 18F-FDG- and 89Zr-panitumumab, negative for both, or positive for one and not the other. The outcome is numbers without dispersion
Time Frame: up to 5 days
Population: Some participants did not have lymph nodes collected, or the collected lymph nodes were not evaluable. Some lymph nodes were not evaluable by all methodologies.
Measure: Number; unit: Lymph Nodes
Units Other Than Participants: Lymph nodes
Groups:
- Tumor-positive Lymph Nodes (by 18F-FDG Scan): Participants whose lymph nodes are positive for cancer.
  Panitumumab-IRDye800: 30 mg administered intravenously (IV)
  Zirconium Zr-89 Panitumumab: 0.8 to 1.2 mCi (29 to 45 Mbq) administered intravenously (IV)
  Pinpoint IR IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  SPY-PHI IR9000 fluorescence imaging system (FIS): Handheld fluorescence-imaging endoscope manufactured by Novadaq
  Explorer Air camera: Fluorescence camera manufactured by SurgVision
  PDE-NEO II camera: Medical infrared camera manufactured by Hamamatsu Photonics KK
  FIS-00 fluorescence imaging system (FIS): Fluorescence imaging system (FIS) manufactured by Hamamatsu Photonics KK
  Da Vinci Firefly Imaging System: Fluorescence-imaging endoscope, mounted or stand-alone, manufactured by Intuitive Surgical Inc
  IGP-ELVIS-v4 Macroscopic Specimen Imager: Macroscopic specimen imager manufactured by LI-COR Biosciences
  Vevo 3100 LAZR-X: Photoacoustic ultrasound imaging system manufactured by VisualSonics
  Pearl Triology Imaging System: Near-infrared fluorescent and bioluminescent imaging system manufactured by LI-COR Biosciences
  Odyssey CLx Imaging System: Infrared fluorescent imaging system manufactured by LI-COR Biosciences
  Leica fluorescence microscope: Fluorescence microscope manufactured by Leica
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
Number analyzed (Participants) | 3 | 5
Number analyzed (Lymph nodes) | 6 | 19
Lymph Nodes
  89Zr-panitumumab-positive & pathology-positive: number analyzed (Lymph nodes) | 5 | 16
  89Zr-panitumumab-positive & pathology-positive | 0 | 4
  89Zr-panitumumab-positive & pathology-negative: number analyzed (Lymph nodes) | 5 | 16
  89Zr-panitumumab-positive & pathology-negative | 0 | 0
  89Zr-panitumumab-negative & pathology-positive: number analyzed (Lymph nodes) | 5 | 16
  89Zr-panitumumab-negative & pathology-positive | 0 | 6
  89Zr-panitumumab-negative & pathology-negative: number analyzed (Lymph nodes) | 5 | 16
  89Zr-panitumumab-negative & pathology-negative | 5 | 6
  18F-FDG-positive & pathology-positive: number analyzed (Lymph nodes) | 6 | 18
  18F-FDG-positive & pathology-positive | 0 | 7
  18F-FDG-positive & pathology-negative: number analyzed (Lymph nodes) | 6 | 18
  18F-FDG-positive & pathology-negative | 0 | 3
  18F-FDG-negative & pathology-positive: number analyzed (Lymph nodes) | 6 | 18
  18F-FDG-negative & pathology-positive | 0 | 2
  18F-FDG-negative & pathology-negative: number analyzed (Lymph nodes) | 6 | 18
  18F-FDG-negative & pathology-negative | 6 | 6
  89Zr-panitumumab-positive & 18F-FDG-positive: number analyzed (Lymph nodes) | 5 | 15
  89Zr-panitumumab-positive & 18F-FDG-positive | 0 | 2
  89Zr-panitumumab-positive & 18F-FDG-negative: number analyzed (Lymph nodes) | 5 | 15
  89Zr-panitumumab-positive & 18F-FDG-negative | 0 | 1
  89Zr-panitumumab-negative & 18F-FDG-positive: number analyzed (Lymph nodes) | 5 | 15
  89Zr-panitumumab-negative & 18F-FDG-positive | 0 | 8
  89Zr-panitumumab-negative & 18F-FDG-negative: number analyzed (Lymph nodes) | 5 | 15
  89Zr-panitumumab-negative & 18F-FDG-negative | 5 | 4

2. Secondary Outcome: Sensitivity and Specificity of 89Zr-panitumumab, 18F-FDG, and Panitumumab-IRDye800
Description: The value of 89Zr-panitumumab and panitumumab-IRDye800 as a label for cancer cells (radiologic or fluorescent, respectively), was assessed by the sensitivity and specificity for the detection of tumor cells in lymph nodes near the tumor. 18F-fluorodeoxyglucose (18F-FDG), an established agent for this use, was also assessed. Sensitivity was assessed as the "true positive rate" of paired measurements, expressed as the proportion (ratio) of the number of specimens positive by histopathology also positive by the test method (test:histopathology). Specificity is the "true negative rate", the proportion of the number of specimens negative by histopathology also negative by the test method. The closer the proportions are to 1, the greater the sensitivity or specificity. The outcome is reported as the sensitivity and specificity of 89Zr-panitumumab, panitumumab-IRDye800, and 18F-fluorodeoxyglucose (18F-FDG). The outcome results are ratios, a number without dispersion.
Time Frame: up to 5 days
Population: Some participants did not have lymph nodes collected, or the collected lymph nodes were not evaluable. Some lymph nodes were not evaluable by all methodologies.Some participants did not have lymph nodes collected, or the collected lymph nodes were not evaluable. Some lymph nodes were not evaluable by all methodologies.
Measure: Number; unit: Ratio
Units Other Than Participants: Lymph nodes
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
Number analyzed (Participants) | 3 | 5
Number analyzed (Lymph nodes) | 6 | 19
Ratio
  89Zr-panitumumab Sensitivity | 0 | 0.4
  89Zr-panitumumab Specificity | 0 | 1.0
  Panitumumab-IRDye800 Sensitivity | 0 | 1.0
  Panitumumab-IRDye800 Specificity Panitumumab-IRDye800 Specificity | 0 | 1.0
  18F-FDG Sensitivity | 0 | 0.78
  18F-FDG Specificity | 0 | 0.67

3. Other Pre Specified Outcome: 89Zr-panitumumab and 18F-FDG False-negatives
Description: The value of experimental 89Zr-panitumumab as a radiologic label was assessed as the number of lymph nodes (LNs) that have false-negative results. A false-negative result in this study is one that does not indicate that cancer is present in the lymph node, when histopathologic evaluation confirms the presence of cancer in the lymph nodes. The outcome is reported as the number of false-negative lymph nodes observed after systemic labeling with 89Zr-panitumumab and 18F-FDG, an established agent for this use. The outcome results are numbers without dispersion.
Time Frame: up to 5 days
Population: as for outcome 1
Measure: Number; unit: Lymph nodes
Units Other Than Participants: Lymph nodes
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
Number analyzed (Participants) | 3 | 5
Number analyzed (Lymph nodes) | 6 | 19
Lymph nodes
  89Zr-panitumumab False-negatives | 0 | 6
  18F-FDG False-negatives | 0 | 2

4. Other Pre Specified Outcome: Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of 89Zr-panitumumab and 18F-FDG
Description: The value of experimental 89Zr-panitumumab as a radiologic label was assessed by determining the positive predictive value (PPV) and the negative predictive value (NPV). PPV is a measure of extent that positive-labeled samples that were actually cancer, expressed as a proportion (ratio) of the number of positive-labeled samples vs samples positive by histopathology (positive label/positive histopathology). NPV is a measure of extent that negative-labeled samples (not positive) that were actually NOT cancer, expressed as a proportion (ratio) of the number of negative-labeled samples vs samples NOT positive by histopathology (negative label/negative histopathology). The closer the proportions are to 1, the better the predictive value. The outcome is reported as the PPV and NPV of 89Zr-panitumumab and 18F-fluorodeoxyglucose (18F-FDG), an established agent for this use. The outcome results are ratios, numbers without dispersion.
Time Frame: up to 5 days
Population: as for outcome 1
Measure: Number; unit: ratio
Units Other Than Participants: Lymph nodes
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
Number analyzed (Participants) | 3 | 5
Number analyzed (Lymph nodes) | 6 | 19
ratio
  89Zr-panitumumab Positive Predictive Value (PPV) | 0 | 0.4
  89Zr-panitumumab Negative Predictive Value (NPV) | 0 | 1.0
  18F-FDG Positive Predictive Value (PPV) | 0 | 0.78
  18F-FDG Negative Predictive Value (NPV) | 0 | 0.67

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Tumor-negative Lymph Nodes (by 18F-FDG Scan) | Tumor-positive Lymph Nodes (by 18F-FDG Scan)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tumor-negative Lymph Nodes (by 18F-FDG Scan) (N=7) | Tumor-positive Lymph Nodes (by 18F-FDG Scan) (N=7)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tumor-negative Lymph Nodes (by 18F-FDG Scan) (N=7) | Tumor-positive Lymph Nodes (by 18F-FDG Scan) (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Other (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Other, hypercarbia (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other, refeeding syndrome, mild (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Other, fistula, nasal-oral, right (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other, - Jackson-Pratt drain with serous drainage and tracheostomy site with mucinous secretion (Surgical and medical procedures) | 0 (0) | 1 (1)
Other, extravasation along anterior abdominal wall consistent with gastrostomy tube leak (Surgical and medical procedures) | 1 (1) | 0 (0)
Other, jejunostomy tube leak (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03733210/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03733210/ICF_002.pdf